CLINICAL TRIAL: NCT00077454
Title: A Phase I Study of Single Agent OSI-774 (Tarceva) (NSC# 718781, IND# 63383) Followed by OSI-774 With Temozolomide for Patients With Selected Recurrent/Refractory Solid Tumors, Including Brain Tumors
Brief Title: Erlotinib and Temozolomide in Treating Young Patients With Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01808; ADVL0214; CDR0000350336; COG-ADVL0214; NCI-04-C-0256; U01CA097452 (NIH); NCT00089934 (obsolete NCT alias)
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Previously Treated Childhood Rhabdomyosarcoma; Recurrent Childhood Brain Tumor; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Malignant Germ Cell Tumor; Recurrent Childhood Medulloblastoma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Neuroblastoma; Recurrent Osteosarcoma
MeSH Terms: conditions — Astrocytoma; Familial ependymoma; Medulloblastoma; Neuroblastoma; Osteosarcoma | interventions — Erlotinib Hydrochloride; Temozolomide

ARMS (1):
- Treatment (erlotinib hydrochloride, temozolomide) (Experimental): Patients receive oral erlotinib once daily on days 1-28. Beginning with course 2, patients also receive oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 23 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Drug: temozolomide; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally (PO)
  Other Names: CP-358,774; erlotinib; OSI-774
Drug: temozolomide — Given PO
  Other Names: SCH 52365; Temodal; Temodar; TMZ
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of erlotinib when given with temozolomide in treating young patients with recurrent or refractory solid tumors. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving erlotinib with temozolomide may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of erlotinib in children with recurrent or refractory solid tumors.

II. Determine the dose-limiting toxic effects of this drug alone and with temozolomide in these patients.

III. Determine the tolerability of this regimen in these patients. IV. Determine the pharmacokinetics of this regimen in these patients.

SECONDARY OBJECTIVES:

I. Determine, preliminarily, the antitumor activity of this regimen in these patients.

OUTLINE: This is a 2-part, multicenter, dose-escalation study of erlotinib. Patients are stratified according to pretreatment (heavily pretreated [received more than 2 prior multiagent myelosuppressive chemotherapy regimens OR received prior craniospinal or pelvic radiotherapy or bone marrow transplantation OR has bone marrow involvement] vs less heavily pretreated).Part 1:

Patients receive oral erlotinib once daily on days 1-28. Beginning with course 2, patients also receive oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 23 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of erlotinib during course 1 only until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Part 2: Patients receive erlotinib (at the MTD) and temozolomide as in part 1.

PROJECTED ACCRUAL: A total of 9-45 patients (9-24 for part 1 and up to 21 for part 2) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* One of the following histologically confirmed solid tumors:

  * Brain tumors
  * Osteogenic sarcoma
  * Rhabdomyosarcoma
  * Soft tissue sarcoma (excluding Ewing's sarcoma)
  * Neuroblastoma
  * Germ cell tumors
* Recurrent or refractory disease
* No known curative therapy exists
* Performance status - Karnofsky 50-100% (for patients age 11 to 21)
* Performance status - Lansky 50-100% (for patients age 10 and under)
* At least 8 weeks
* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3 (transfusion independent*)
* Hemoglobin > 8.0 g/dL (transfusion allowed)
* Bilirubin < 1.5 times upper limit of normal (ULN)
* ALT < 2.5 times ULN
* Albumin ≥ 2 g/dL
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min
* Creatinine based on age as follows:

  * ≤ 0.8 mg/dL for patients age 5 and under
  * ≤ 1.0 mg/dL for patients 6 to 10
  * ≤ 1.2 mg/dL for patients 11 to 15
  * ≤ 1.5 mg/dL for patients age 15 to 21
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow tablets (for patients in part 2 only)
* No uncontrolled infection
* Recovered from all prior immunotherapy
* At least 7 days since prior biologic therapy
* At least 3 months since prior stem cell transplantation and no evidence of active graft-versus-host disease
* More than 1 week since prior growth factors
* No concurrent prophylactic growth factor therapy
* No concurrent immunotherapy
* No concurrent biologic therapy
* More than 2 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and recovered
* No other concurrent chemotherapy
* No concurrent systemic corticosteroids except for treatment of increased intracranial pressure or symptomatic tumor edema in patients with CNS tumors

  * No concurrent steroids as an antiemetic
* Concurrent dexamethasone for patients with CNS tumors allowed provided patient has been on a stable or decreasing dose for at least 1 week before study entry
* Recovered from all prior radiotherapy
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 6 weeks since prior substantial bone marrow irradiation
* At least 6 months since prior craniospinal radiotherapy
* At least 6 months since prior radiotherapy to 50% or more of the pelvis
* At least 8 weeks since prior standard-fraction radiotherapy for patients with recurrent brain tumors unless there is biopsy proof of recurrent tumor
* Prior radiosurgery within the past 9 months allowed provided there is documentation of progressive disease by biopsy, positron-emission tomography (PET) scan, or MR spectroscopy
* No concurrent radiotherapy
* More than 1 week since prior CYP3A4 inhibitors
* More than 4 weeks since prior CYP3A4 inducers
* More than 5 days since prior proton-pump inhibitors
* More than 2 days since prior H_2 blockers
* No prior erlotinib
* No concurrent enzyme-inducing anticonvulsants
* No concurrent proton-pump inhibitors
* No concurrent H2 blockers
* No other concurrent investigational agents
* Concurrent antacids allowed provided the antacid is not administered 2 hours before, during, and 2 hours after erlotinib administration

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2004-02; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | 56 days (2 courses)
Maximum-tolerated dose (MTD) based on the incidence of DLT as assessed by NCI CTCAE version 3.0 | 56 days (2 courses)
Pharmacokinetics of erlotinib hydrochloride | At baseline and at 0.5, 1, 2, 4, 6, 8, and 24 hours of course 1

CONTACTS AND LOCATIONS:
Overall Officials: Regina Jakacki, Principal Investigator — COG Phase I Consortium
Locations (1):
- COG Phase I Consortium, Arcadia, California, United States